CLINICAL TRIAL: NCT00175266
Title: Islet Transplantation in Type 1 Diabetic Patients Using Campath-1H and Infliximab Induction
Brief Title: Islet Transplantation Using Campath-1H and Infliximab Induction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3516
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Type 1 Diabetes
Keywords: islet; transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Alemtuzumab; Infliximab

INTERVENTIONS:
Drug: alemtuzumab
Procedure: islet transplant
Drug: infliximab

SUMMARY:
Islet transplantation has been investigated as a treatment for Type 1 diabetes mellitus in selected patients with inadequate glucose control despite insulin therapy. However, the perennial hope that such an approach would result in long-term freedom from the need for exogenous insulin, with stabilization of the secondary complications of diabetes, has failed to materialize in practice. The goal of the present study is therefore to improve the safety and efficacy of clinical islet-alone transplantation by minimizing dependence on calcineurin-inhibitor therapy - thereby avoiding potential nephrotoxicity, and furthermore improving success with single-donor islet infusions by avoiding all diabetogenic immunosuppression. Campath-1H, combined with Infliximab induction therapy provides a unique opportunity to minimize dosing of maintenance long-term immunosuppression while further promoting islet engraftment.

DETAILED DESCRIPTION:
This is a single-centre, prospective, open-label study in Type 1 diabetic participants receiving an islet cell transplant; all participants will receive Campath-1H + Infliximab induction therapy followed by sirolimus and ultra-low dose tacrolimus maintenance therapy.

The primary objective of this protocol is to assess the safety of this treatment regimen in adult Type 1 diabetic participants receiving their first islet transplant.

ELIGIBILITY:
Inclusion Criteria:

* must have Type 1 diabetes mellitus for more than 5 years
* diabetes must be complicated by at least one of the following situations that persist despite intensive insulin management efforts. The complicating situations are (1) Reduced awareness of hypoglycemia, as defined by the absence of adequate autonomic symptoms at plasma glucose levels of < 3.0 mmol/L; (2) Metabolic lability/instability, characterized by MAGE ≥ 11.0 mmol/L and wide swings in blood glucose despite optimal diabetes therapy; and (3) Despite efforts at optimal glucose control, progressive secondary complications of diabetes, including retinopathy, neuropathy, or nephropathy

Exclusion Criteria:

* Severe co-existing cardiac disease
* Active alcohol or substance abuse
* Psychiatric disorder making the subject not a suitable candidate for transplantation
* Active infection including hepatitis C, hepatitis B, HIV, or TB
* Any history of or current malignancies except squamous or basal skin cancer
* BMI > 28 kg/m2 or body weight > 85 kg at screening visit
* Positive fasting C-peptide response on assessment (2 positive results)
* Creatinine clearance < 80 mL/min/1.73 m2
* Serum creatinine > 150 µmol/L
* Macroalbuminuria (urinary albumin excretion rate > 300 mg/24h)
* Baseline Hb < 105g/L in women, or < 130 g/L in men
* Baseline LFT's outside of normal range
* Untreated proliferative retinopathy
* Positive pregnancy test, intent for future pregnancy or male subjects' intent to procreate, failure to follow effective contraceptive measures, or presently breast feeding
* Previous transplant, or evidence of sensitization on PRA
* Insulin requirement > 1.0 IU/kg/day
* HbA1C > 0.12
* Hyperlipidemia (fasting LDL cholesterol > 3.4 mmol/L, treated or untreated; and/or fasting triglycerides > 2.3 mmol/L)
* Under treatment for a medical condition requiring chronic use of steroids
* Use of coumadin or other anticoagulant therapy (except aspirin) or subject with PT INR > 1.5
* Untreated Addison's disease
* Untreated Celiac disease
* Untreated thyroid disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12

CONTACTS AND LOCATIONS:
Overall Officials: A.M. James Shapiro, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta - Clinical Islet Transplant Program, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Gala-Lopez B, Kin T, O'Gorman D, Pepper AR, Senior P, Humar A, Shapiro AM. Microbial contamination of clinical islet transplant preparations is associated with very low risk of infection. Diabetes Technol Ther. 2013 Apr;15(4):323-7. doi: 10.1089/dia.2012.0297. Epub 2013 Feb 25. PMID 23438305